CLINICAL TRIAL: NCT07257809
Title: A Multicenter, Single-arm Exploratory Clinical Study Evaluating the Efficacy and Safety of T-DM1 in Patients With Breast Cancer Who Developed Thrombocytopenia.
Brief Title: Herombopag Treated T-DM1 Induced Platelet Reduction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yinduo Zeng, chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQBP-IIT-2025
Record Dates: First submitted 2025-09-03; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A (Experimental): Herombopag， initial dose 7.5 mg po qd d1-14
  Interventions: Drug: Herombopag Olamine Tablets

INTERVENTIONS:
Drug: Herombopag Olamine Tablets — Herombopag 7.5 mg po qd，d1-14

SUMMARY:
This is a single-arm study planned to enroll 56 breast cancer patients who experienced grade 2 or higher thrombocytopenia following prior chemotherapy and achieved normalization (platelet count ≥100 × 109/L and ≥200 × 109/L) through intervention.

ELIGIBILITY:
Inclusion：

* Age 18-75 years, any gender;
* Pathologically diagnosed with breast cancer based on histological or cytological examination, and previously treated with neoadjuvant anti-HER-2 therapy followed by T-DM1 adjuvant therapy;
* Experienced grade 2 or higher tumor treatment-related thrombocytopenia during the previous T-DM1 treatment cycle, with platelet count restored to ≥100 × 109/L and ≤200 × 109/L prior to the next treatment;
* ECOG performance status score: 0-2;
* Planned to undergo at least two additional treatment cycles including T-DM1 administration, with the dose of T-DM1 in the current cycle consistent with the previous cycle;
* Expected survival of ≥12 weeks and able to tolerate the current treatment regimen for at least two cycles or more;
* Expected to have good compliance, able to follow up on treatment efficacy and adverse reactions as required by the protocol.

Exclusion:

* A history of other malignant tumors diagnosed within the past 3 years;
* Patients with mental or neurological disorders who are unable to cooperate;
* Patients who are scheduled to undergo or have previously undergone organ or bone marrow transplantation;
* Patients with hematopoietic system disorders other than chemotherapy-induced thrombocytopenia (CTIT), including but not limited to leukemia, primary immune thrombocytopenia, myeloproliferative disorders, multiple myeloma, and myelodysplastic syndrome;
* Patients with a history of any arterial or venous thrombotic events within the past 6 months prior to screening;
* Severe bleeding manifestations within 2 weeks prior to screening, such as gastrointestinal or central nervous system bleeding;
* Participation in a clinical trial of the same type of drug within 4 weeks prior to enrollment;
* Pregnant or lactating women;
* Patients with a history of hypersensitivity to the study drug;
* Patients deemed ineligible by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 56 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2027-09-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of grade I thrombocytopenia according to CTCAE4.0 | From enrollment to the end of treatment at 6 weeks
  The proportion of patients with platelet counts <100 × 109/L according to CTCAE4.0

SECONDARY OUTCOMES:
the proportion of salvage platelet transfusion therapy | From enrollment to the end of treatment at 6 weeks
  Proportion of patients requiring platelet transfusion therapy during treatment
time to platelet counts ≥100 × 109/L | From enrollment to the end of treatment at 6 weeks
  Median time to achieve and maintain platelet counts ≥100 × 109/L from the start of Hetrombopag until the next treatment cycle;
Proportion of T-DM1with unexpected administration | From enrollment to the end of treatment at 6 weeks
  Proportion of patients who experienced delay, dose reduction, or discontinuation of T-DM1 due to thrombocytopenia
proportion of adverse events | From enrollment to the end of treatment at 6 weeks
  According to CTC AE 4.0 to evaluate profile of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yinduo Zeng, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China